CLINICAL TRIAL: NCT07000955
Title: Tolerance and Pharmacokinetic/Pharmacokinetic Study of IBI362 15mg Administered Multiple Times in Chinese Patients With Moderate to Severe Obesity
Brief Title: Tolerance and Pharmacokinetic/Pharmacokinetic Study of IBI362 15mg in Patients With Moderate to Severe Obesity
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CIBI362B104
Record Dates: First submitted 2025-05-08; First posted 2025-06-03 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Tirzepatide; mazdutide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: blinded: participant, investigator, outcome assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IBI362 (Experimental): Stage 1: subcutaneous injection, qw; dose ranging from 2.0mg to 15.0mg，44w Stage 2: subcutaneous injection, q2w; 12.0mg or 15.0mg, 12w;
  Interventions: Drug: IBI362
- Placebo (Placebo Comparator): Stage 1: subcutaneous injection, 0mg, qw, 44w Stage 2: subcutaneous injection, dose ranging from 2.0mg to 6.0mg，qw, 12w
  Interventions: Drug: Placebo
- Tirzepatide (Active Comparator): Open label: subcutaneous injection, qw, dose ranging from 2.5mg to 15.0mg, 44w
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Tirzepatide — Tirzepatide administered subcutaneously (SC) once a week.
  Arms: Tirzepatide
Drug: Placebo — Placebo administered subcutaneously (SC) once a week.
  Arms: Placebo
Drug: IBI362 — IBI362 administered subcutaneously (SC) once a week.
  Arms: IBI362

SUMMARY:
This study is a multicenter, randomized, partially double-blind (double-blind in both the IBI362 group and the placebo group, with the tirbopeptide group open), placebo and active drug controlled design study

ELIGIBILITY:
Inclusion Criteria:

* 1. The age at the time of screening is 18 to 55 years old (including both ends), male or female;
* 2. BMI≥32.5 kg/m2 during screening;
* 3. At the time of screening, after simple diet and exercise control for at least 12 weeks, the weight change was less than 5% [(Maximum weight within 3 months before screening - minimum weight within 3 months before screening)/maximum weight within 3 months before screening ×100%, self-reported by the subjects]
* 4. Fertile subjects agreed to take the contraceptive measures stipulated in this protocol throughout the study and within 3 months after the last treatment. Female subjects with reproductive capacity must have negative pregnancy test results during screening. Female subjects should not breastfeed throughout the study and within 3 months after the last treatment;
* 5. Voluntarily sign the informed consent form and be willing to strictly abide by the requirements and restrictions in the informed consent form and protocol throughout the research period, including but not limited to: diet, exercise, lifestyle management, planned injection of research drugs, keeping research diaries, and completing relevant questionnaires, etc;

Exclusion Criteria:

* 1. The investigator suspected that the subjects might be allergic to the study drug or component or have an allergic constitution;
* 2. Use any of the following drugs or treatments within 3 months before screening including but not limited to GLP-1R, GIPR, GCGR, any drugs, Chinese herbal medicines, health supplements or meal replacements that have an impact on body weight, or participated in other clinical trials;
* 3. There is a history or evidence of any of the following diseases before screening or at the time of screening including but not limited to diabetes, have received or plan to undergo bariatric surgery during the research period in the past, with retinopathy in the past or at the time of screening, secondary diseases or drugs lead to obesity, have a history of depression in the past or have a history of serious mental illness in the past, hypertension that has not been stably controlled at the time of screening after at least 4 weeks of antihypertensive drug treatment, a history of malignant tumors was present during the screening, heart disease, A 2A or 2B history or family history of medullary thyroid carcinoma and multiple endocrine adenomatosis (MEN) , history of acute and chronic pancreatitis, limb deformity or disability, have a history of suicidal tendencies or suicidal behaviors, etc according to the protocol.
* 4. Any of the laboratory examination indicators meets the following standards during screening: serum calcitonin ≥20ng/L during screening, alanine aminotransferase ≥2.0×ULN and/or aspartate aminotransferase ≥2.0×ULN and/or total bilirubin ≥1.5×ULN and/or alkaline phosphatase ≥2.0×ULN, eGFR is less than 60 Ml/min/1.73 m2, abnormal thyroid function including FT3, FT4, or TSH, fasting triglycerides ≥5.64 mmol/L (500 mg/dl), blood amylase or lipase 1.0 x ULN;
* 5. During the screening, the 12-lead electrocardiogram showed a heart rate of <50 beats per minute or >90 beats per minute;
* 6. There were clinically significant ECGs abnormalities during the screening;
* 7. History of other risk factors for tachycardia;
* 8. The blood donation volume and/or blood loss volume within 3 months prior to screening is ≥400mL, or bone marrow donation has been performed, or there are anemia-related diseases such as hemoglobinopathy, hemolytic anemia, sickle cell anemia, etc., or hemoglobin.. 110g/ L (male) or 100g/L (females).
* 9. The investigators believe that the subjects have any other factors that may affect the efficacy or safety evaluation of this study and are not suitable to participate in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2025-06-17 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-05-14 (Estimated)

PRIMARY OUTCOMES:
The Incidence of adverse events and serious adverse events during the treatment period | week 44
The suicidal ideation and behavior of subjects evaluated by Columbia-Suicide Severity Rating Scale (C-SSRS) | week 44
The incidence rates of Adverse Event of Special Interest | week 44
The value of systolic and diastolic pressures | week 44
The RR interval, PR interval, heart rate, QT interval, Fridericia-corrected QT interval, and any abnormal reporting results of 12-lead electrocardiogram | week 44
Any adverse event evaluated by laboratory examinations | week 44
  Including amylase, lipase, alanine aminotransferase [ALT], aspartate aminotransferase [AST], calcitonin, urinary albumin-to-creatinine ratio [UACR], creatine kinase [CK], lactate dehydrogenase [LDH], etc
The value of pulse rate | week 44

SECONDARY OUTCOMES:
Evaluate the pharmacokinetic (PK) characteristics of IBI362 | week 44
  Maximum Plasma Concentration Area under the concentration-time curve
The change in body weight from baseline | week 44
Immunogenicity | week 44
  The incidence of serum anti-IBI362 antibody (ADA) and neutralizing antibody (Nab)
The change in waist circumference from baseline | week 44
Changes and percentage changes of abdominal visceral fat (VAT) content, abdominal subcutaneous fat (SAT) content, and abdominal total fat (TAAT) content relative to the baseline | week 44
Changes and percentage changes of liver fat content compared with the baseline | week 44
The changes in insulin resistance index (HOMA2-IR) and islet β-cell function index (HOMA2-B) from baseline calculated by the concentration of fasting blood glucose and the concentration of fasting insulin | week 44
The change in body-mass index from baseline | week 44
The change in neck circumference from baseline | week 44
The change in hip circumference from baseline | week 44
The change in waist circumference/hip circumference ratio from baseline | week 44
Changes in hemoglobin A1c (HbA1c%) , from baseline | week 44
Changes in fasting blood glucose , from baseline | week 44
Changes in Fasting insulin, from baseline | week 44
Changes in Fasting C-peptide, from baseline | week 44

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China